CLINICAL TRIAL: NCT07211724
Title: Methamphetamine Use Disorder Support in Heart Failure (Meth HF) Pilot Study
Brief Title: Methamphetamine Use Disorder Support in Heart Failure Pilot Study
Acronym: Meth-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Los Angeles General Medical Center (Other)
Responsible Party: Principal Investigator, Tien Ng, Professor of Clinical Pharmacy and Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-25-00064
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Methamphetamine Use Disorder
Keywords: Heart Failure; Methamphetamine use disorder; Meth-associated cardiomyopathy; Multidisciplinary
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Multidisciplinary HF clinic integrating MUD management (Other): This is a single-arm study to evaluate the feasibility and preliminary efficacy of a multidisciplinary HF clinic which integrates MUD management along with standard-of-care guideline directed HF management.
  Interventions: Other: MUD Management (contingency management +/- adjunctive MUD pharmacotherapy); Other: HF GDMT management

INTERVENTIONS:
Other: MUD Management (contingency management +/- adjunctive MUD pharmacotherapy) — Management of MUD will be individualized for each study patient. All patients will receive behavioral counseling utilizing motivational interviewing and education and offered a contingency management (CM) plan incentivizing abstinence from meth. Several pharmacotherapies are recommended for the treatment of MUD: mirtazapine, bupropion and naltrexone, or bupropion monotherapy. If required, adjunctive MUD pharmacotherapy will be added to the CM guided by comorbid conditions, patient characteristics, and characteristics of use.
Other: HF GDMT management — As per standard clinical care, patients will be followed by a cardiologist for HF management including assessment for GDMT optimization.

SUMMARY:
Heart failure (HF) affects over 6 million people in the US and is a major cause of both hospital admissions and death. HF has many causes and contributing factors. One of the most aggressive forms of HF is associated with methamphetamine abuse, which has become its own epidemic in the US over the past twenty years. People who use methamphetamine tend to develop HF at a much younger age, with more severe disease and more serious consequences. A recent analysis using nationwide data, methamphetamine use doubled the risk of death or hospitalizations compared to non-users in patients with HF. Thus, methamphetamine users with HF represent a very high-risk group of patients from a healthcare perspective.

HF may be reversible in some patients who use methamphetamine if patients can achieve 1) abstain from further methamphetamine use and 2) consistently take all the medications that can improve HF. These two goals are very difficult to achieve in practice, as the care of both methamphetamine addiction and HF requires specialized medical expertise and intensive regular follow up of patients. In general, achievement of one goal is not possible without the other. Patients who use methamphetamine have poor adherence to medical follow-up and therapies, and abstinence from methamphetamine is difficult to maintain. This is further complicated because the current model of HF care does not incorporate treatment for methamphetamine use.

The current study proposes to launch a multidisciplinary clinic that treats both HF and methamphetamine use disorder at the same time. The HF care will be led by a cardiologist while the methamphetamine use treatment will be led by a psychiatric clinical pharmacist trained in addiction medicine. State-of-the-art HF care will include optimization of four pillar HF medications. Methamphetamine use treatment will include counseling and incentivized abstinence known as contingency management (CM). The investigators will manage the patients in the clinic for 6 months total.

The investigators are interested in demonstrating that this integrated clinic model will result in improved delivery of care for these patients by reporting the rates of successful abstinence from methamphetamine, improved optimization of the four HF medications, and enhanced patient reported quality of life over the 6 months of follow up. The investigators will also collect data on the costs associated with providing this level of care and estimate a range of potential cost-savings.

DETAILED DESCRIPTION:
Prospective, open-label, single-arm study to evaluate the feasibility and preliminary efficacy of a multidisciplinary HF clinic which integrates MUD management along with standard-of-care guideline directed HF management. The MUD treatment plan will be pragmatic, consisting of behavioral counseling, CM with or without pharmacotherapy (see below). Patients with HF and concomitant active meth use will be enrolled consecutively and managed in the clinic for 6 months. The pragmatic approach to MUD treatment will allow for individualization of therapy plans reflecting current MUD guidelines. The overarching objective of the current proposal is to demonstrate the feasibility and preliminary value of a HF clinic for meth users that integrates MUD treatment. The central hypothesis is that incorporation of simultaneous meth use abstinence incentives and aid with HF management in a singular clinic visit model will improve care delivery metrics associated with improved HF outcomes. The hypothesis aligns with HF guidelines that emphasize the essential role of incorporating comorbidity management into routine care of patients with HF.

Specific Aim 1 will define the rate of successful abstinence from meth with implementation of a multidisciplinary meth HF clinic utilizing contingency +/- pharmacologic management strategies alongside standard HF care in a prospective, open-label pragmatic study. Patients with HF and documented meth use will be consecutively enrolled for follow-up in the study clinic. Along with standard-of-care management of HF, patients will work with the addiction medicine pharmacist to receive an individualized MUD treatment plan for 6 months. Implementation of an effective MUD treatment plan will result in both improved abstinence from meth, as well as adherence to clinic visits and HF therapies over the 6 months of follow-up, establishing the feasibility and model for this multidisciplinary integrated clinic.

Specific Aim 2 will assess the clinical value of the meth HF clinic to improve HF care quality metrics. As a pilot study, patient adherence to HF GDMT and follow-up appointments will be descriptively quantified, along with achievement of GDMT target doses at 1, 3, and 6 months. Changes in patient quality of life from baseline will be ascertained utilizing the Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Since MUD represents an established barrier to patient adherence with medical therapies, the integration of MUD with HF care will improve these HF care quality metrics associated with improved patient outcomes in HF. These data will demonstrate the preliminary value for this multidisciplinary integrated clinic.

Specific Aim 3 will enumerate the healthcare resources and costs required for implementation, and further attempt to estimate the range of cost savings associated with the meth HF clinic. To demonstrate feasibility and replicability, the costs associated with this care model will be estimated through prospective collection of care delivery data across all study patients, including personnel time and other direct costs of the MUD treatment. Cost savings will be estimated based on projected reductions in health resource use (e.g., reduced out- and inpatient encounters). The cost and savings components will be the foundation for designing both a payer-perspective budget impact analysis, and a societal-perspective full cost-effectiveness analysis for incorporation into a future randomized, controlled study of the clinical and economic impacts of the clinic.

The study will establish the feasibility and preliminary value of an innovative model of care delivery for very high-risk patients with HF and MUD that reduces barriers to optimizing the care and benefit. The broader impact will be established by demonstrating that increased meth abstinence improves adherence and GDMT optimization, underscoring the value of systems that provide a holistic patient-centric approach to HF management. Specifically, the achievement of many of the guideline-recommended HF clinical performance and quality measures can be enhanced by incorporating SUD treatment into the standard of care for HF.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure diagnosis meeting universal definition criteria with left ventricular ejection fraction ≤ 40%
* Active methamphetamine use and stated desire to cease (confirmed by patient self-reported history of active use and /or positive urine toxicology obtained as part of routine patient care); physician verifying patients meets criteria for MUD.
* Age 18 years or older
* Empaneled to LA General Medical Center/DHS
* Able to provide informed consent (translated consent forms will be used for non-English speakers)

Exclusion Criteria:

* Polysubstance use (excluding tobacco and marijuana)
* Documented history of alcohol use disorder (DSM-5) or alcohol dependence (ICD-11). Intermittent alcohol use below these thresholds (e.g. social use) is not an exclusion.
* Cardiogenic shock requiring mechanical circulatory support at time of presentation
* Acute coronary syndrome, acute pulmonary embolism, or hemodynamically significant arrhythmia on admission
* Pregnancy
* Acute psychiatric condition requiring immediate treatment or significantly impairing their ability to provide informed consent or participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence from Methamphetamine | From enrollment to the end of intervention at 6 months
  The rate of abstinence from meth will be defined as the percentage of negative urine toxicology results/number of visits. A total of 36 visits/person to the Heart Failure clinic over the 6 months of follow-up will be scheduled.
GDMT optimization - drug class prescribing | From enrollment to the end of intervention at 6 months
  Guideline-directed medical therapies (GDMT) optimization will be evaluated by % prescribed all 4 GDMT drug classes
GDMT optimization - dosing | From enrollment to the end of intervention at 6 months
  Guideline-directed medical therapies (GDMT) optimization will be evaluated by % of patients on GDMT target doses and half-target doses.

SECONDARY OUTCOMES:
BSCS score changes over time | From enrollment to the end of intervention at 6 months
  A Brief Substance Craving Scale (BSCS) is a 4-item Likert-scale patient-reported tool that measures frequency and intensity of cravings. Scores range from 0-12, with higher scores indicating greater craving. Survey will be conducted at last visit of each month in a total of 6 months.
KCCQ-12 score changes over time | From enrollment to the end of intervention at 6 months
  A 12-item Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated tool and performance measure for quality of care, assessing patient symptoms, functional limitations, and quality of life in patients with HF. Scores range from 0-100, with higher scores indicating better health status. Survey will be conducted at last visit of each month in a total of 6 months.

OTHER OUTCOMES:
Health care costs | From enrollment to the end of intervention at 6 months
  Enumerate the healthcare resources and costs required for implementation, and further attempt to estimate the range of cost savings associated with the meth HF clinic. To demonstrate feasibility and replicability, the costs associated with this care model will be estimated through prospective collection of care delivery data across all study patients, including personnel time and other direct costs of the MUD treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tien Ng, PharmD, Principal Investigator — University of Southern California, Alfred E. Mann School of Pharmacy and Pharmaceutical Sciences
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - University of Southern California, Alfred E. Mann School of Pharmacy and Pharmaceutical Sciences, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozkurt B, Coats AJS, Tsutsui H, Abdelhamid CM, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Michael Felker G, Filippatos G, Fiuzat M, Fonarow GC, Gomez-Mesa JE, Heidenreich P, Imamura T, Jankowska EA, Januzzi J, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, Seferovic P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal definition and classification of heart failure: a report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure: Endorsed by the Canadian Heart Failure Society, Heart Failure Association of India, Cardiac Society of Australia and New Zealand, and Chinese Heart Failure Association. Eur J Heart Fail. 2021 Mar;23(3):352-380. doi: 10.1002/ejhf.2115. Epub 2021 Mar 3. PMID 33605000
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Wu JR, Moser DK. Medication Adherence Mediates the Relationship Between Heart Failure Symptoms and Cardiac Event-Free Survival in Patients With Heart Failure. J Cardiovasc Nurs. 2018 Jan/Feb;33(1):40-46. doi: 10.1097/JCN.0000000000000427. PMID 28591004
- [Background] Gandhi S, Mosleh W, Sharma UC, Demers C, Farkouh ME, Schwalm JD. Multidisciplinary Heart Failure Clinics Are Associated With Lower Heart Failure Hospitalization and Mortality: Systematic Review and Meta-analysis. Can J Cardiol. 2017 Oct;33(10):1237-1244. doi: 10.1016/j.cjca.2017.05.011. Epub 2017 May 24. PMID 28807523
- [Background] Douglass AR, Maister A, Moeller KE, Salwan A, Vallabh A, Waters K, Payne GH. Exploring the harm reduction paradigm: the role of Board-Certified Psychiatric Pharmacists. Ment Health Clin. 2024 Aug 2;14(4):253-266. doi: 10.9740/mhc.2024.08.253. eCollection 2024 Aug. PMID 39104432
- [Background] Clinical Guideline Committee (CGC) Members; ASAM Team; AAAP Team; IRETA Team. The ASAM/AAAP Clinical Practice Guideline on the Management of Stimulant Use Disorder. J Addict Med. 2024 May-Jun 01;18(1S Suppl 1):1-56. doi: 10.1097/ADM.0000000000001299. PMID 38669101
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Reddy PKV, Ng TMH, Oh EE, Moady G, Elkayam U. Clinical Characteristics and Management of Methamphetamine-Associated Cardiomyopathy: State-of-the-Art Review. J Am Heart Assoc. 2020 Jun 2;9(11):e016704. doi: 10.1161/JAHA.120.016704. Epub 2020 May 29. PMID 32468897
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Zhao SX, Deluna A, Kelsey K, Wang C, Swaminathan A, Staniec A, Crawford MH. Socioeconomic Burden of Rising Methamphetamine-Associated Heart Failure Hospitalizations in California From 2008 to 2018. Circ Cardiovasc Qual Outcomes. 2021 Jul;14(7):e007638. doi: 10.1161/CIRCOUTCOMES.120.007638. Epub 2021 Jul 13. PMID 34256572
- See also: Center for Behavioral Health Statistics and Quality SAaMHSA. Substance Abuse and Mental Health Services Administration. Key Substance Use and Mental Health Indicators in the United States: Results from the 2018 National Survey on Drug Use and Health. — https://www.samhsa.gov/data/sites/default/files/cbhsq-reports/NSDUHNationalFindingsReport2018/NSDUHNationalFindingsReport2018.pdf